CLINICAL TRIAL: NCT00086411
Title: Comparing Smoking Treatment Programs for Lighter Smokers
Brief Title: Comparing Smoking Treatment Programs for Lighter Smokers - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-15365-1; R01DA015365 (NIH)
Record Dates: First submitted 2004-07-01; First posted 2004-07-07 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Tobacco Use Disorder
Keywords: light smokers, smoking cessation treatment programs
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine; Bupropion; Medication Therapy Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: Bup+MM (Experimental): bupropion and MM counseling with placebo patch
  Interventions: Drug: bupropion; Behavioral: Medication Management; Drug: placebo patch
- 2 Bup+Mayo (Experimental): bupropion and Mayo counseling with placebo patch.
  Interventions: Drug: bupropion; Behavioral: Mayo Counseling; Drug: placebo patch
- 3 Patch+MM (Placebo Comparator): patch and MM counseling with placebo pills
  Interventions: Drug: nicotine transdermal system; Behavioral: Medication Management; Drug: placebo bupropion
- 4 Patch+Mayo (Experimental): patch and Mayo counseling with placebo pills
  Interventions: Drug: nicotine transdermal system; Behavioral: Mayo Counseling; Drug: placebo bupropion

INTERVENTIONS:
Drug: nicotine transdermal system — starting with 21 or 14mg dependent on number of cigarettes per day smoked upon entry in the study; titrated down over 8 weeks.
  Other Names: Nicoderm
  Arms: 3 Patch+MM; 4 Patch+Mayo
Drug: bupropion — 150 mg/day X 3 days 300mg/day for 60 days Total 9 weeks
  Other Names: Zyban
  Arms: 1: Bup+MM; 2 Bup+Mayo
Behavioral: Medication Management — Brief manual based therapy; four 15 minute session over 10 weeks.
  Arms: 1: Bup+MM; 3 Patch+MM
Behavioral: Mayo Counseling — Manual based therapy; Weekly 30 minute sessions for 10 weeks
  Arms: 2 Bup+Mayo; 4 Patch+Mayo
Drug: placebo patch — placebo patch containing no nicotine
  Arms: 1: Bup+MM; 2 Bup+Mayo
Drug: placebo bupropion — placebo pills
  Arms: 3 Patch+MM; 4 Patch+Mayo

SUMMARY:
The purpose of this study was to compare two different types of Food and Drug Administration (FDA) approved smoking cessation medications (nicotine patch or bupropion) used in conjunction with two levels of counseling. It was hypothesized that the higher level of counseling would have the highest rates of treatment completion and highest rates of abstinence.

DETAILED DESCRIPTION:
The study compared a minimal level counseling model to a higher level counseling model plus one of two types of FDA approved smoking cessation products (bupropion or the nicotine patch)used to achieve long term abstinence among lighter smokers. Each participant received both products under blinded conditions meaning that neither the participant nor the counselor knew which product was real or a placebo. The primary goal was to determine the combination or combinations of high or low intensity counseling and pharmacotherapy (either bupropion or the nicotine patch) that were most effective for lighter smokers. The main hypothesis was that higher level counseling would contribute to improved outcomes meaning that more counseling would be associated higher abstinence rates following the completion of treatment and at longer term follow-up.

ELIGIBILITY:
Light smokers (6-15 cigarettes per day

Inclusion Criteria:

Mentally and physically stable, non-pregnant, light smokers (6-15 cigarettes per day)

Exclusion Criteria:

Please contact site for more information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Gariti, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Gariti P, Levin S, Whittingham T, Barou D, Kampman KM, Lynch K, Halbert CH, Alterman A. Why do those who request smoking treatment fail to attend the first appointment? J Subst Abuse Treat. 2008 Jul;35(1):62-7. doi: 10.1016/j.jsat.2007.08.009. Epub 2007 Oct 10. PMID 17931823
- [Result] Gariti P, Lynch K, Alterman A, Kampman K, Xie H, Varillo K. Comparing smoking treatment programs for lighter smokers with and without a history of heavier smoking. J Subst Abuse Treat. 2009 Oct;37(3):247-55. doi: 10.1016/j.jsat.2009.01.006. Epub 2009 Mar 31. PMID 19339135
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample consists of 260 self-referred lighter smokers to an urban university setting. The first participant was enrolled in February 2005, and the last follow-up was completed in March 2008. A total of 302 met confirmatory screening criteria, and 260 were enrolled.
Pre-assignment Details: An in-person confirmatory screening interview consisted of a medical examination, structured psychological interview (Mini International Neuropsychiatric Interview; Sheenan et al., 1997), and biochemical testing (i.e., carbon monoxide reading of expired air [CO], blood alcohol concentration,and urine drug test).
Groups:
- 1 Bup+MM: bupropion and MM with placebo patch
- 3 Patch+MM: patch and MM with placebo pills
- 4 Patch+Mayo: patch and Mayo counseling with placebo patch
Period: Overall Study
Arm/Group | 1 Bup+MM | 2 Bup+Mayo | 3 Patch+MM | 4 Patch+Mayo
Started | 70 | 63 | 62 | 65
Completed | 59 | 52 | 49 | 53
Not Completed | 11 | 11 | 13 | 12
Not completed — Lost to Follow-up | 11 | 11 | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- 1: Bup+MM: bupropion and MM with placebo patch
- Total: Total of all reporting groups
Arm/Group | 1: Bup+MM | 2 Bup+Mayo | 3 Patch+MM | 4 Patch+Mayo | Total
Number analyzed (Participants) | 70 | 63 | 62 | 65 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.5) | 42.4 (12.6) | 45.8 (12.6) | 43.1 (11.3) | 43.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 31 | 35 | 38 | 148
  Male | 26 | 32 | 27 | 27 | 112
Region of Enrollment [Number; unit: participants]
  United States | 70 | 63 | 62 | 65 | 260

OUTCOME MEASURES:

1. Primary Outcome: Percent Treatment Sessions Attended
Description: Completion of Treatment and Smoking Cessation by Two Different Types of Medications and Counseling Types at 12, 26, and 52 Weeks Post-treatment Initiation. The counseling types were Medication Management (MM) and Mayo counseling models. MM counseling was a 4 session lower intensity counseling model and Mayo counseling was a 10 session higher intensity model.
  A twofold definition of treatment completion included both medication and counseling session adherence. Treatment completion was defined as consistently taking the active medication as prescribed (80%) of the time during the medication period and attending at least 7 of the 10 required High C sessions or 3 of the 4 Low C sessions. Participants had to meet both requirements to be designated as full treatment completers.
  Seven-day point prevalence abstinence was the primary measure of abstinence at follow-up Weeks 12, 24, and 52. Abstinence was confirmed by biochemical testing.
Time Frame: 52 weeks
Measure: Mean (Standard Error); unit: Percentage of attended tx. sessions
Arm/Group | 1: Bup+MM | 2 Bup+Mayo | 3 Patch+mm | 4 Patch+Mayo
Number analyzed (Participants) | 70 | 63 | 62 | 65
Percentage of attended tx. sessions | 77.9 (.05) | 85.9 (.04) | 66.8 (.06) | 66.6 (.06)
Statistical Analysis 1: Comparison: 1: Bup+MM vs 2 Bup+Mayo vs 3 Patch+mm vs 4 Patch+Mayo; Rates of abstinence were addressed using a generalized estimating equations (GEE) logistic regression model. Counseling type and medication type were entered as the main explanatory variables along with time and the interaction of these factors, together with some covariates (described below). The sample size provided 80% power to detect a difference of about 14% between groups across three time points (i.e., 12, 26, and 52 weeks post-treatment initiation; Test type: Superiority or Other; p < 0.017, GEE model for repeated binary outcomes — The p-value was adjusted for multiple comparisons; Model included hx of heavy smoking, elevated depression, cigarettes per day, gender, and race; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.77 to 2.25], Standard Error of Mean 0.2734 — The above was for the main effect of BUP versus NTX on cessation

2. Secondary Outcome: Delineate Mediators Associated With Different Treatment Conditions (i.e., Medication Compliance, Participant Views of Self-help Written Materials and Counseling Type.
Time Frame: 52 weeks
Population: PI is no longer with institution. All efforts have been exhausted to locate this data, but no data is available to be reported
Arm/Group | 1: Bup+MM | 2 Bup+Mayo | 3 Patch+MM | 4 Patch+Mayo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The reported time frame for study related serious adverse events was 1 year. Two participants died prior to the week 52 follow-up of non-study related problems. The reported time frame for adverse events is the first 12 weeks (3 weeks post medication).
Arm/Group | 1: Bup+MM | 2 Bup+Mayo | 3 Patch+mm | 4 Patch+Mayo
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/63 | 1/62 | 0/65
Other Adverse Events (participants affected / at risk) | 1/70 | 3/63 | 0/62 | 2/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1: Bup+MM (N=70) | 2 Bup+Mayo (N=63) | 3 Patch+mm (N=62) | 4 Patch+Mayo (N=65)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Bup+MM (N=70) | 2 Bup+Mayo (N=63) | 3 Patch+mm (N=62) | 4 Patch+Mayo (N=65)
Medication stopped due to reported side effects. (General disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Missing data from some early terminations from treatment (i.e., 2 or less visits) may reflect dissatisfaction with counseling assignment or medication effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes